CLINICAL TRIAL: NCT01354847
Title: Influence of Extracorporeal Circulation on Platelet Function of Patients Undergoing Cardiac Surgery - a Prospective Observational Study
Brief Title: Influence of Extracorporeal Circulation on Platelet Function of Patients Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Christian F. Weber, MD, Dr. Dr. Christian Friedrich Weber, Goethe University
Other Study IDs: MEAECC
Record Dates: First submitted 2011-05-02; First posted 2011-05-17 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Acquired Platelet Function Disorder
Keywords: extracorporeal circulation; platelet dysfunction; Multiplate electrode aggregometry analyses; Multiplate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiac surgery patients: cardiac surgery patients scheduled for elective complex cardiac surgery
  Interventions: Device: Multiple electrode aggregometry analyses (Multiple Electrode Aggregometry, Multiplate(R), Verum Diagnostica, Munich, Germany)

INTERVENTIONS:
Device: Multiple electrode aggregometry analyses (Multiple Electrode Aggregometry, Multiplate(R), Verum Diagnostica, Munich, Germany) — ex vivo platelet aggregation at several intraoperative and postoperative measuring points.

SUMMARY:
This study is planned to investigate the relationship between duration of extracorporeal circulation and the extent of (acquired) platelet dysfunctions in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Patients undergoing complex cardiac surgery are planned to be included. At several intra- and postoperative measuring point, blood is drawn for multiple electrode aggregometry to investigate ex-vivo platelet aggregation as a surrogate for platelet function.

Transfusion rate of allogenic blood products as well as postoperative blood loss is planned to be recorded.

ELIGIBILITY:
Inclusion Criteria:

* duration of extracorporeal circulation > 120 min

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac surgery patients undergoing complex cardiac surgery (double valve, aortic surgery, combined - or redo procedures)
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Changes in arachidonic acid induced platelet aggregation as compared to baseline (before extracorporeal circulation) | Baseline (before extracorporeal circulation) and 60, 90, 120, 150 and 180 minutes after extracorporal circulation as well as ad admission to ICU
  Multiple Electrode aggregometry parameters

SECONDARY OUTCOMES:
Changes in Adenosin Diphosphate (ADP) and Thrombin induced platelet aggregation as compared to baseline (before extracorporeal circulation) | Baseline (before extracorporeal circulation) and 60, 90, 120, 150 and 180 minutes after extracorporal circulation as well as ad admission to ICU
  Multiple electrode aggregometry analyses

CONTACTS AND LOCATIONS:
Overall Officials: Christian F Weber, M.D., Principal Investigator — Goethe University Frankfurt, Theodor Stern Kai 7, 60590 Frankfurt, Germany; Christian Reyher, M.D., Study Chair — Goethe University Frankfurt, Clinic for Anesthesiology, Theodor Stern Kai 7, 60590 Frankfurt, Germany
Locations (1):
- Goethe - University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Velik-Salchner C, Maier S, Innerhofer P, Kolbitsch C, Streif W, Mittermayr M, Praxmarer M, Fries D. An assessment of cardiopulmonary bypass-induced changes in platelet function using whole blood and classical light transmission aggregometry: the results of a pilot study. Anesth Analg. 2009 Jun;108(6):1747-54. doi: 10.1213/ane.0b013e3181a198ac. PMID 19448196